CLINICAL TRIAL: NCT03144310
Title: TO EVALUATE THE ROLE OF LUNG ULTRASONOGRAPHY FOR DETECTION OF ATELECTASIS IN ADULTS UNDERGOING ROBOT ASSISTED LAPAROSCOPIC PELVIC SURGERIES
Brief Title: To Evaluate the Role of Lung Ultrasonography for Detection of Atlelectasis in Robot Assisted Laproscopic Pelvic Sugeries
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Rahul Kathuria, junior resident doctor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/3067/MD/320
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: to Detect the Incidence of Atelectasis
MeSH Terms: interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: lung ultrasound — lung ultrasound and blood gas
  Other Names: blood gas analysis

SUMMARY:
Pre op ultrasound with chest auscultation and arterial blood gas, after extubation ultrasound with chest auscultation and blood gas, 12hrs chest auscultation with ultasaound, 24 hrs chest auscultation and ultrasound to see atelectasis

DETAILED DESCRIPTION:
Pre op ultrasound with chest auscultation and arterial blood gas, after extubation ultrasound with chest auscultation and blood gas, 12hrs chest auscultation with ultasaound, 24 hrs chest auscultation and ultrasound to see atelectasis inclusion criteria: age 18 to 70 yrs age ASA I and II robot assisted pelvic surgeries in steep trendelenburg position

exclusion criteria: cardiac disese severe obstructive and restrictive disease upper airways infection ASAIII and IV

ELIGIBILITY:
Inclusion Criteria:

* ASA Iand II age 18-70 yrs robot assisted pelvis surgeries

Exclusion Criteria:

* ASA II and IV cardiac and lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA Iand II age 18-70 yrs
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
incidence of atelectasis | 24hrs
  incidence of atelectasis in adults after extubation undergoing robot assisted pelvic laproscopic surgery in steep trendelenberg position using ultrasound

SECONDARY OUTCOMES:
risk factor identification | 24hrs
  risk factor identification of post operative atelectasis

CONTACTS AND LOCATIONS:
Overall Officials: Pgimer, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: No